CLINICAL TRIAL: NCT00527111
Title: A Randomized Phase II Trial of Pre-operative Chemoradiotherapy With or Without Cetuximab (ERBITUX(R)) in Locally-advanced Adenocarcinoma of the Rectum
Brief Title: Pre-op Rectal ChemoRad +/- Cetuximab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Oncology Research (Industry)
Collaborators: Bristol-Myers Squibb (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05102; CA225269 (Other: Bristol-Myers-Squibb)
Record Dates: First submitted 2007-09-07; First posted 2007-09-10 (Estimated); Results first posted 2016-11-03 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-09

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Cetuximab; Fluorouracil; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chemoradiotherapy plus Cetuximab (Experimental): Pelvic irradiation plus 5-fluorouracil plus cetuximab
  Interventions: Drug: Cetuximab; Drug: 5-fluorouracil; Radiation: Pelvic irradiation
- Chemoradiotherapy alone (Active Comparator): Pelvic irradiation plus 5-fluorouracil
  Interventions: Drug: 5-fluorouracil; Radiation: Pelvic irradiation

INTERVENTIONS:
Drug: Cetuximab
  Other Names: Erbitux
  Arms: Chemoradiotherapy plus Cetuximab
Drug: 5-fluorouracil
  Other Names: 5-FU
Radiation: Pelvic irradiation
  Other Names: Radiotherapy

SUMMARY:
The purpose of this research study is to find out what effects (good and bad) cetuximab has on rectal cancer.

DETAILED DESCRIPTION:
Rectal cancer remains a significant cause of morbidity and mortality in the United States. Standard treatment for patients with locally advanced rectal cancer generally includes combined chemotherapy and radiotherapy administered either before (neoadjuvant) or after (adjuvant) definitive surgical resection. Published data from Germany has suggested advantages to a neoadjuvant strategy. Currently, the standard concurrent chemoradiotherapy regimen in the United States is pelvic irradiation administered concurrently with 5-fluorouracil (5-FU) given as a protracted venous infusion. However, local recurrence remains a problem. Recently completed randomized trials of chemoradiotherapy have demonstrated local recurrence rates between 8-17% even with currently accepted standard chemoradiotherapy and adequate surgical management.

Several recent trials have explored the use of radiotherapy and cetuximab with good results.

Because of the non-overlapping toxicity profiles and the potentially diverse and complimentary mechanisms of action, the combination of chemotherapy plus ERBITUX given concurrently with pelvic radiotherapy may improve on the outcomes seen with current standards for patients with locally advanced adenocarcinoma of the rectum.

ELIGIBILITY:
Inclusion Criteria:

Note: Please see Section 8.1 for the necessary "Prestudy Assessments".

A patient will be eligible for inclusion in this study if s/he meets all of the following criteria:

* Has a histologically confirmed diagnosis of newly diagnosed adenocarcinoma of the rectum (tumor within 15 cm of the anal verge). Location of tumor (lower 1/3rd vs. middle or upper 1/3rd) and pre-treatment nodal status (N0 vs. N1 or N2) will be recorded in the eCRF. Patients with only non-measurable disease are eligible as long as they meet the other disease requirements in this criterion as well as all other eligibility criteria.
* Has tumor that is locally advanced (T3/T4 or lymph node positive) by preoperative assessment with CT or MRI imaging or transrectal ultrasonography.
* Has no evidence of distant metastases by radiographic staging
* Has an ECOG Performance Status (PS) 0-1
* Is greater than 18 years of age
* Has adequate marrow and organ system function as assessed by the following lab values:

White blood cell (WBC) count See protocol for specific details Absolute neutrophil count (ANC) See protocol for specific details Hemoglobin See protocol for specific details Total bilirubin See protocol for specific details AST and ALT See protocol for specific details Serum creatinine See protocol for specific details Platelet count See protocol for specific details

* Sexually active women of childbearing potential must use an effective method of birth control during the course of the study, in a manner such that risk of failure is minimized.

Prior to study enrollment, women of childbearing potential (WOCBP) must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy. In addition, men enrolled on this study should understand the risks to any sexual partner of childbearing potential and should practice an effective method of birth control.

All WOCBP MUST have a negative pregnancy test within 3 weeks prior to registration (confirmed within 7 days prior to first receiving investigational product). If the pregnancy test is positive, the patient must not receive investigational product and must not be enrolled in the study.

In addition, all WOCBP should be instructed to contact the Investigator immediately if they suspect they might be pregnant (eg, missed or late menstrual period) at any time during study participation.

The Investigator must immediately notify BMS in the event of a confirmed pregnancy in a patient participating in the study.

* Has signed a Patient Informed Consent Form
* Has signed a Patient Authorization Form

Exclusion Criteria:

* A patient will be excluded from this study if s/he meets any of the following criteria:
* Has another disease similar to one being studied (ie, colon cancer)
* Has evidence of distant metastases by radiographic staging
* Has had prior treatment for the current disease
* Has had prior stem cell or bone marrow transplant or any organ transplant with the exception of corneal transplant or cadaver bone graft
* Has a history of hypersensitivity to any of study treatments
* Has had a prior severe infusion reaction to a monoclonal antibody
* Has received prior therapy, at any time, which specifically and directly targets the EGFR pathway
* Has a significant history of uncontrolled cardiac disease; ie, uncontrolled hypertension, unstable angina, recent myocardial infarction (within prior 6 months), uncontrolled congestive heart failure, or cardiomyopathy with decreased ejection fraction
* Has evidence of CNS involvement (CNS imaging is not required for study enrollment unless clinically suspected CNS disease is present.)
* Has a serious uncontrolled intercurrent medical or psychiatric illness, including serious infection or Gilbert's Syndrome
* Has a history of other malignancy within the last 5 years (except cured basal cell carcinoma of skin and carcinoma in situ of uterine cervix), which could affect the diagnosis or assessment of any of the study drugs. Patients, who have received prior radiotherapy to any regional site other than the pelvis, as long as all other inclusion criteria are met, could be considered for enrollment after discussion with Dr. McCollum.
* Is a pregnant or nursing woman
* Is unable to comply with requirements of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2007-02; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D McCollum, MD, Principal Investigator — US Oncology Research
Locations (41):
- United States (41):
  - Oncology Associates D.B.A. Hematology Oncology Physicians & Extenders, Tucson, Arizona
  - Melbourne Internal Medicine Associates, Melbourne, Florida
  - Advanced Medical Specialties, Miami, Florida
  - Cancer Centers of Florida, P.A., Ocoee, Florida
  - Cancer Care & Hematology Specialists of Chicagoland, PC, Niles, Illinois
  - Central Indiana Cancer Centers, Indianapolis, Indiana
  - Kansas City Cancer Centers-Southwest, Overland Park, Kansas
  - Alliance Hematology Oncology PA, Westminster, Maryland
  - Missouri Cance Associates, Columbia, Missouri
  - St. Joseph Oncology, Inc., Saint Joseph, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - New York Oncology Hematology, P.C., Albany, New York
  - Cancer Centers of North Carolina, Raleigh, North Carolina
  - Willamette Valley Cancer Center, Eugene, Oregon
  - Texas Oncology - Amarillo, Amarillo, Texas
  - Texas Oncology Cance Center, Austin, Texas
  - Mamie McFaddin Ward Cancer Center, Beaumont, Texas
  - Texas Cancer Center at Medical City, Dallas, Texas
  - Methodist Charlton Cancer Ctr., Dallas, Texas
  - Texas Oncology, P.A., Dallas, Texas
  - Texas Cancer Center, Denton, Texas
  - El Paso Cancer Treatment Ctr, El Paso, Texas
  - Texas Oncology, P.A., Fort Worth, Texas
  - Lake Vista Cancer Center, Lewisville, Texas
  - Longview Cance Center, Longview, Texas
  - Allison Cancer Center, Midland, Texas
  - Texas Oncology-Odessa, Odessa, Texas
  - Paris Regional Cancer Center, Paris, Texas
  - HOAST - Medical Dr., San Antonio, Texas
  - Texas Cancer Center - Sherman, Sherman, Texas
  - Texas Oncology Cancer Center-Sugar Land, Sugar Land, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Texas Oncology Cancer Care and Research, Waco, Texas
  - Texas Oncology, P.A., Webster, Texas
  - Texoma Cancer Center, Wichita Falls, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Highline Medical Oncology, Burien, Washington
  - Cancer Care Northwest-South, Spokane, Washington
  - Northwest Cancer Specialists-Vancouver, Vancouver, Washington
  - Yakima Valley Mem Hosp/North Star Lodge, Yakima, Washington
  - Raleigh Regional Cancer Center, Beckley, West Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemoradiotherapy Plus Cetuximab: Pelvic irradiation plus 5-fluorouracil plus cetuximab
  Cetuximab
  5-fluorouracil
  Pelvic irradiation
- Chemoradiotherapy Alone: Pelvic irradiation plus 5-fluorouracil
  5-fluorouracil
  Pelvic irradiation
Period: Overall Study
Arm/Group | Chemoradiotherapy Plus Cetuximab | Chemoradiotherapy Alone
Started | 70 | 69
Completed | 50 | 47
Not Completed | 20 | 22
Not completed — Adverse Event | 14 | 13
Not completed — Death | 0 | 1
Not completed — Investigator Request | 2 | 1
Not completed — Patient Request | 2 | 5
Not completed — Other | 2 | 2

BASELINE CHARACTERISTICS:
Population: ITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemoradiotherapy Plus Cetuximab | Chemoradiotherapy Alone | Total
Number analyzed (Participants) | 70 | 69 | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (11.0) | 61.4 (11.7) | 58.6 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 21 | 47
  Male | 44 | 48 | 92
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 59 | 60 | 119
  Black | 8 | 4 | 12
  Hispanic | 1 | 3 | 4
  Asian | 2 | 1 | 3
  Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 70 | 69 | 139

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Pathologic Response Rate (pCR) With 95% Confidence Interval.
Description: A pathologic complete response (pCR) is defined as no pathologic evidence of invasive disease at the primary site in the bowel wall or in examined mesorectal tissue and/or lymph nodes.
Time Frame: 5 years
Population: Post surgery population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemoradiotherapy Plus Cetuximab | Chemoradiotherapy Alone
Number analyzed (Participants) | 64 | 60
percentage of participants | 26.6 [16.3 to 39.1] | 26.7 [16.1 to 39.7]

2. Secondary Outcome: To Determine Objective Response Rate (ORR) Based on RECIST Local Recurrence-free Survival in These Patient Groups; Overall and Recurrence-free Survival in These Cohorts.
Description: Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of the LD of target lesions taking as reference the baseline sum LD.
Time Frame: 5 years
Population: Evaluable Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemoradiotherapy Plus Cetuximab | Chemoradiotherapy Alone
Number analyzed (Participants) | 67 | 62
percentage of participants | 52.2 [39.7 to 64.6] | 43.5 [31.0 to 56.7]

3. Secondary Outcome: 5- Year Overall Survival (OS) Rate
Description: Overall survival is measured from the date of randomization to the date of death for a dead patient. If a patient is still alive or is lost to follow up, the patient will be censored at the date of last contact.
Time Frame: 5 years
Population: ITT population
Measure: Number (95% Confidence Interval); unit: probability of overall survival
Arm/Group | Chemoradiotherapy Plus Cetuximab | Chemoradiotherapy Alone
Number analyzed (Participants) | 70 | 69
probability of overall survival | 0.81 [0.69 to 0.89] | 0.68 [0.53 to 0.79]

4. Secondary Outcome: Recurrence-free Survival (RFS) Rate at 5 Years
Description: RFS is measured from the date of randomization to the date of first documented disease recurrence or date of death, whichever comes first. If a patient neither recurrences nor dies, this patient will be censored at the date of last contact.
Time Frame: 5 years
Population: ITT population
Measure: Number (95% Confidence Interval); unit: probability of recurrence-free survival
Arm/Group | Chemoradiotherapy Plus Cetuximab | Chemoradiotherapy Alone
Number analyzed (Participants) | 70 | 69
probability of recurrence-free survival | 0.65 [0.51 to 0.76] | 0.585 [0.44 to 0.71]

5. Secondary Outcome: KRAS Mutation Rate
Description: Percentage of Participants with KRAS mutation.
Time Frame: 5 years
Population: ITT population with KRAS test
Measure: Number; unit: percentage of participants with mutation
Arm/Group | Chemoradiotherapy Plus Cetuximab | Chemoradiotherapy Alone
Number analyzed (Participants) | 40 | 34
percentage of participants with mutation | 32.5 | 44.0

ADVERSE EVENTS:
Time Frame: During the whole treatment period, up to 30 days following last dose.
Description: For treatment patients only, assessed at each treatment visit.
Arm/Group | Chemoradiotherapy Plus Cetuximab | Chemoradiotherapy Alone
Serious Adverse Events (participants affected / at risk) | 10/67 | 5/62
Other Adverse Events (participants affected / at risk) | 61/67 | 47/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemoradiotherapy Plus Cetuximab (N=67) | Chemoradiotherapy Alone (N=62)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 1 (1)
COLITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
DEHYDRATION (Gastrointestinal disorders) | 5 (5) | 2 (2)
DIARRHEA (Gastrointestinal disorders) | 5 (5) | 1 (2)
ENTERITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
FEVER (General disorders) | 1 (1) | 0 (0)
MUCOSITIS (Infections and infestations) | 1 (1) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 2 (3) | 0 (0)
SWALLOWING PAINFUL (Gastrointestinal disorders) | 0 (0) | 1 (1)
TACHYCARDIA ATRIAL (Cardiac disorders) | 1 (1) | 0 (0)
VOLUME BLOOD DECREASED (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
WEAKNESS GENERALIZED (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemoradiotherapy Plus Cetuximab (N=67) | Chemoradiotherapy Alone (N=62)
ABDOMINAL PAIN (Gastrointestinal disorders) | 5 (6) | 8 (8)
ANEMIA (Blood and lymphatic system disorders) | 5 (6) | 6 (8)
ANOREXIA (Gastrointestinal disorders) | 16 (19) | 13 (15)
CHILLS (General disorders) | 7 (7) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 8 (9) | 5 (5)
DEHYDRATION (Gastrointestinal disorders) | 7 (8) | 8 (13)
DIARRHEA (Gastrointestinal disorders) | 36 (67) | 33 (60)
DRY SKIN (Skin and subcutaneous tissue disorders) | 5 (6) | 0 (0)
FEVER (General disorders) | 6 (6) | 0 (0)
HAND-FOOT SYNDROME (Skin and subcutaneous tissue disorders) | 2 (4) | 9 (14)
HEADACHE (General disorders) | 13 (14) | 1 (1)
HYPOKALEMIA (Metabolism and nutrition disorders) | 7 (11) | 1 (1)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 10 (15) | 4 (4)
LEUCOPENIA (Blood and lymphatic system disorders) | 4 (4) | 5 (10)
MUCOSAL SORES (Infections and infestations) | 4 (5) | 5 (5)
MUCOSITIS (Infections and infestations) | 19 (25) | 12 (21)
MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 2 (3) | 4 (5)
NAUSEA (Gastrointestinal disorders) | 18 (22) | 13 (22)
NEUTROPENIA (Blood and lymphatic system disorders) | 5 (6) | 4 (7)
PAIN (General disorders) | 3 (4) | 6 (6)
RASH (Skin and subcutaneous tissue disorders) | 50 (99) | 5 (5)
STOMATITIS (Gastrointestinal disorders) | 5 (6) | 5 (6)
VOMITING (Gastrointestinal disorders) | 6 (7) | 5 (7)
WEAKNESS (General disorders) | 25 (31) | 19 (20)
WEIGHT LOSS (General disorders) | 7 (8) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No